CLINICAL TRIAL: NCT02446639
Title: Assessment the Dosage of Troponin T Hypersensitive Dosage in a Patient Population Hemodialysis and Peritoneal Dialysis (ECHOTnT)
Brief Title: Assessment the Dosage of Troponin T Hypersensitive Dosage in a Patient Population Hemodialysis and Peritoneal Dialysis
Acronym: ECHOTnT
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC13_0056
Record Dates: First submitted 2015-04-28; First posted 2015-05-18 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Renal Failure Chronic Requiring Dialysis
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Blood collection

SUMMARY:
"Troponin T (TnT) is a component of the contractile apparatus of the striated musculature. Although the function of TnT is the same in all striated muscles found in the heart to form a TNT (cardiac TnT) differing significantly TnT of the skeletal muscles. Because of its high tissue specificity, cardiac TnT is a specific marker and highly sensitive of myocardial injury.

Asymptomatic elevations of troponins is frequently found in patients with chronic renal failure in stage V, which present no clinical signs of acute or electrical myocardial injury.

Many studies have been conducted in recent years to explain the origin and clinical significance of this elevation, but the results are controversial: cardiac dysfunction, left ventricular hypertrophy or chronic inflammation.

Besides the effect of the dialysis session was evaluated on this biological parameter in different studies which together do not find Impact hemodialysis session on the value of troponin Achieving dosages rate hypersensitive serum troponin T in a dialysis population, will:

* to determine the evolution of TnT in time and what are the characteristics of the patients for whom this rate varies
* to know what its evolution during the session,
* to identify if possible the criteria that are responsible for the variation in the direction of increasing and / or its reduction
* and to characterize patients whose base rate is higher than the 99 percentile in the absence of clinical symptoms which could lead to establish reference population for this specific normal values. The Purpose of this study is to evaluate the serum troponin T in a hypersensitive dialysis population and verify what is the influence of the hemodialysis session, the session parameters and intradialytic events on changes in serum troponin T hypersensitive after a hemodialysis session. "

DETAILED DESCRIPTION:
Current care study, single-center, uncontrolled, no randomised, open and prospective.

Two hundred fifty patients on hemodialysis and / or peritoneal dialysis for more than 3 months may be included in the study for a total period of 7 months.

Hemodialysis patients will be informed at the weekly routine visits. Regarding peritoneal dialysis patients, a meeting can be organized with the physician. And the oral agreement of the patient will be collected during a second visit or meeting.

The protocol provides four follow-up visits: at baseline, 4 weeks, 12 and 24 weeks.

During these visits, the patient will have a clinical examination and a measure of the serum troponin T. Blood samples are realized in the usual conditions of the center - for hemodialysis patients: midweek as instructed by the usual protocol of the center. - for peritoneal dialysis patients: when the monthly routine consultation.

ELIGIBILITY:
Inclusion Criteria:

* Patient in Hemodialysis and/or peritoneal dialysis for more than 3 months
* Major patient
* Patient who can express his consent
* Collection of the not opposition
* Affiliated to the national insurance scheme

Exclusion Criteria:

* Encircled woman
* Patients in poor condition general or whose likely survival does not exceed 6 months
* Patient presenting an evolutionary acute pathology or a neoplastic disease
* Patient with significant cardiac problems
* Rhabdomyolysis known muscular disease and active
* Patient presenting an unchecked active infection,HIV
* Patient included in another protocol of search which could interfere with the objectives of this study
* Patient psychiatric or incapable to give an informed consent or to pursue the study.
* Minor Patient
* Under guardianship patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing haemodialysis or peritoneal dialysis for more than 3 months
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
To assess serum troponin T in a hypersensitive dialysis population | At the time of the inclusion
  Assessment of serum troponin T hypersensitive measured just before the second dialysis week (at the time of inclusion).

SECONDARY OUTCOMES:
To estimate the influence of the session of haemodialysis | At the time of the inclusion
  For the patients in haemodialysis, measures of the serum troponin before and after dialysis
To estimate the evolution of the serum Troponin T | At the time of the inclusion, at 4 weeks, at 12 weeks and at 24 weeks
  measures of the serum troponin T before dialysis
To compare the measures of serum troponin T between the patients diabetics and the patients not diabetics, between the patients with cardiac histories and the patients without histories | At the time of the inclusion
  Clinical questionnaire
To compare the evolution of the measures of the serum Troponin T between the patients having undergone one cardiac event and the patients not having presented cardiac events | At the time of the inclusion, at 4 weeks, at 12 weeks and at 24 weeks
  Clinical questionnaire
To compare the measures of the serum Troponin T according to the technique of dialysis: Hemodialysis versus peritoneal dialysis. | At the time of the inclusion
  Clinical questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Centre ECHO, Rezé, France